CLINICAL TRIAL: NCT02911519
Title: Efficacy of a Brief Group Psychoeducation Program Aimed at Patients With Schizophrenia and Their Families: A Clinical Controlled Trial
Brief Title: Brief Group Psychoeducation for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salud Mental Integral S.A.S. (Other)
Collaborators: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAM001
Record Dates: First submitted 2016-09-19; First posted 2016-09-22 (Estimated); Results first posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Patient Education
MeSH Terms: conditions — Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Group Psychoeducation (Experimental): It was designed after a review of the literature on the subject; content and procedures will be written in a manual. They will be five sessions of two hours once a week. Each session will be conducted by a clinical psychologist and a general practitioner trained in group management.
  Interventions: Other: Brief Group Psychoeducation; Other: Treatment as Usual
- Treatment as Usual Only (Active Comparator): The patients in both arms of the intervention will receive this type of attention. The TAU is the psychiatric care that patients with schizophrenia usually receive in the clinic. The frequency of consultations varies depending on severity of symptoms usually split between one and six months.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Other: Brief Group Psychoeducation — First session: describe the clinical manifestations of schizophrenia, deny myths, and inform on the biological nature of the disorder. Second session: provide updated information regarding pharmacological treatment, their side effects and the importance of adherence to treatment. Third session: Achieving recognition of personal responsibility for the lifestyle, routine, physical care and the risk of addiction; awareness of the importance of self-monitoring of symptoms and the development of cognitive, behavioral and emotional strategies. Fourth Session: To recognize the role of family members in the treatment, the problem of expressed emotions and communication in times of crisis. Fifth Session: To know the rights and duties of patients and their families in the current health care system.
  Arms: Brief Group Psychoeducation
Other: Treatment as Usual — The patients in both arms of the intervention will receive this type of attention. The TAU is the psychiatric care that patients with schizophrenia usually receive in the clinic. This is done in consultation of 30 minutes, in which the psychiatrist evaluates the clinical condition of the patient and psychosocial factors that may be affecting, prescribes drugs according to protocols and clinical care and answers questions about the disorder. In the consultation a brochure with information is given about schizophrenia. The frequency of consultations varies depending on severity of symptoms usually split between one and six months.

SUMMARY:
This study evaluates the addition of psychoeducation to treatment as usual in the treatment of adults with schizophrenia for relapse prevention. Half of participants will receive a brief (5 sessions) psychoeducation intervention and treatment as usual in combination, while the other half will receive treatment as usual only.

DETAILED DESCRIPTION:
Schizophrenia is a chronic persistent and disabling psychiatric syndrome whose primary feature is the presence of delusions, hallucinations, disorganized speech or behavior, catatonic behavior and negative symptoms (poverty of thought, social isolation, decreased expression of emotions and motivation for activities). Its incidence in one year is 15.9 per 100,000 inhabitants; its prevalence is 4.3 per 1,000 inhabitants and has been shown to be more common among men, migrant population, urban area, developed countries and greater latitude. It is associated with: 1) Increased mortality rates compared to the general population 2) Disability is one of the top ten causes of years lived with disability in people between 15 and 44 years old, which can be explained by incomplete remission of up to 80% of affected patients and psychotic relapses (5-7). 3) High economic costs given by relapses, hospitalizations, decreased labor productivity and financial and emotional burden for families (8,9). The latter has increased in the last 50 years by changes in the mental health care systems throughout the world that have left families a greater responsibility in caring for patients so they would need more knowledge about the disorder, treatment and rehabilitation (10,11). All this justifies the search for strategies aimed at preventing psychosis crisis increase the period between crises and decrease disability (12,13,14). Psychoeducation is one of the strategies that have been raised so far (15).

Psychoeducation is an intervention based on the structured and systematic knowledge acquisition of a mental disorder, with the aim of improving their clinical prognosis and reduce care costs (15,16,17). There are various designs of psychoeducative programs, they can be individual or group, involving only patients, family or both, or short (less than 10 sessions) or longer. There is insufficient evidence to establish whether any of these methods is most effective, and with respect to the psychoeducation in general, available studies suggest that it may have beneficial effect on reduction in relapses, adherence, hospital stay, global functioning and quality of life (19). However, these studies have methodological limitations such as lack of clarity in the generation and concealment of randomized allocation sequence, non-blind assessment of outcomes and frequent losses in monitoring, suggesting that the effects observed for psychoeducation may not be valid and could be overestimated. Additionally, the cultural characteristics and health system of each country may limit the applicability of studies, which may be necessary to evaluate the efficacy in sites with particular conditions (20).

In a private psychiatric clinic in Medellin primarily serving patients who belong to the contributory scheme of health care, Brief Psychoeducation Group Program was designed (five sessions) for Patients with Schizophrenia and their Families (PGSF). It was decided to include both patients and relatives because some studies suggest there may be advantages and generally patients with this disorder should go out accompanied. It will be group because some authors have argued that it could have more benefits than individual, to facilitate meetings with others, by facilitating the encounter with other people with similar conditions, which could have additional therapeutic effects and be more cost-effective (19). It will be five sessions because it was considered that they could cover the main issues and ensure the attendance at all sessions, taking into account the economic conditions and time restrictions most for most relatives. It is very important to evaluate the effectiveness of this program because that will allow making informed decisions regarding the implementation in this and other psychiatric care institutions in the country. In addition, there are not any controlled clinical trials in Colombia that evaluate the effectiveness of a psychoeducational intervention for this disorder.

Therefore, the research question is: In a psychiatric clinic of Medellin (Colombia), What is the effectiveness of a Brief Psychoeducational Group Program for Patients with Schizophrenia and their Families (PGSF) added to their Outpatient Treatment as Usual (TAU) compared with TAU to reduce the risk of relapse?

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia according to the International Classification of Diseases in its tenth edition (ICD-10).
2. The relative who attend the PGSF must have lived with the patient in the last year and is preferred to be their primary caregiver.
3. Agree to participate in the investigation.

Exclusion Criteria:

1. Be involved in another group psychoeducation program.
2. Have clinically significant psychotic symptoms that indicate "decompensation" with a score in the Clinical Global Impressions Scale for severity (CGI-S) 3 or greater.
3. Dementia.
4. Moderate mental retardation
5. Drug Addiction. (Consumption of active illegal psychoactive substances or alcohol during the last three months.
6. Medical comorbidity whose life expectancy is less than one year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny G Valencia, M.D. M.Sc. Ph.D., Principal Investigator — Salud Mental Integral - Samein - SAS

IPD SHARING:
Plan to Share IPD: Yes
The information will be available at the sponsor webpage.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were selected from the users who attended ambulatory control in the Comprehensive Mental Health Clinic that serves Colombian health care users. Through telephone call and referral by treating psychiatrists, those users who, due to clinical history, were diagnosed with schizophrenia, were invited to participate.
Groups:
- Brief Group Psychoeducation: Brief Group Psychoeducation: First session: describe the clinical manifestations of schizophrenia, deny myths, and inform on the biological nature of the disorder. Second session: provide updated information regarding pharmacological treatment, their side effects and the importance of adherence to treatment. Third session: Achieving recognition of personal responsibility for the lifestyle, routine, physical care and the risk of addiction; awareness of the importance of self-monitoring of symptoms and the development of cognitive, behavioral and emotional strategies. Fourth Session: To recognize the role of family members in the treatment, the problem of expressed emotions and communication in times of crisis. Fifth Session: inform duties and rights of the patient and his family in the Colombian health system and administrative procedures related to patient care.
  This Brief Group Psychoeducation also received Treatment as Usual.
- Treatment as Usual Only: The patients in both arms of the intervention received this type of attention. The TAU is the psychiatric care that patients with schizophrenia usually receive in the clinic.
  Treatment as Usual: The TAU is the psychiatric care that patients with schizophrenia usually receive in the clinic. This is done in consultation of 30 minutes, in which the psychiatrist evaluates the clinical condition of the patient and psychosocial factors that may be affecting, prescribes drugs according to protocols and clinical care and answers questions about the disorder. In the consultation a brochure with information is given about schizophrenia. The frequency of consultations varies depending on severity of symptoms usually split between one and six months.
Period: Overall Study
Arm/Group | Brief Group Psychoeducation | Treatment as Usual Only
Started | 90 | 86
Completed | 88 | 82
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 2
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Group Psychoeducation | Treatment as Usual Only | Total
Number analyzed (Participants) | 90 | 86 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 90 | 86 | 176
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 51
  Male | 62 | 63 | 125
Marital Status [Count of Participants; unit: Participants]
  Single | 70 | 69 | 139
  Civil Union/Married | 12 | 13 | 25
  Divorced/Widow | 8 | 4 | 12
Employment [Count of Participants; unit: Participants]
  Employed | 35 | 30 | 65
  Unemployed | 55 | 56 | 111
Age of onset [Median (Inter-Quartile Range); unit: years] | 22.5 [17.7 to 33.0] | 20.0 [16.0 to 28.0] | 22.0 [17.0 to 30.0]
Duration of disorder [Median (Inter-Quartile Range); unit: years] | 16.5 [5.0 to 27.0] | 16.0 [8.7 to 27.0] | 16.0 [7.0 to 27.0]
Number of episodes [Median (Inter-Quartile Range); unit: psychotic episodes] — Number of psychotic episodes of each patient before the intervention
  psychotic episodes | 3.0 [1.7 to 7.2] | 3.5 [2.0 to 7.2] | 3.0 [2.0 to 7.0]
Number of hospitalizations [Median (Inter-Quartile Range); unit: Number of hospitalizations] — Number of hospitalizations of each patient before the intervention
  Number of hospitalizations | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 5.0] | 2.0 [1.0 to 4.0]
The Clinical Global Impression - Severity scale (CGI-S) [Median (Inter-Quartile Range); unit: units on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. The score is between 1 and 7 in which 1 is normal and 7 represents the most extremely ill patients
  units on a scale | 3.0 [2.0 to 3.0] | 3.0 [2.0 to 3.0] | 3.0 [2.0 to 3.0]
Scale for the Assessment of Positive Symptoms (SAPS) [Median (Inter-Quartile Range); unit: units on a scale] — The Scale for the Assessment of Positive Symptoms (SAPS) is a rating scale to measure positive symptoms in schizophrenia. SAPS is split into 4 domains, and within each domain separate symptoms are rated from 0 (absent) to 5 (severe). The score is between 0 and 155, a higher score on the scale represents a worse clinical status.
  units on a scale | 19.0 [4.7 to 31.2] | 11.0 [4.0 to 24.0] | 14.0 [4.0 to 28.5]
Scale for the Assessment of Negative Symptoms (SANS) [Median (Inter-Quartile Range); unit: units on a scale] — The Scale for the Assessment of Negative Symptoms (SANS) is a rating scale to measure negative symptoms in schizophrenia. The scale is between 0 and 95. The higher score represents worse clinical status.
  units on a scale | 36.0 [18.7 to 52.0] | 33.5 [23.7 to 53.3] | 34.5 [21.0 to 52.0]
Schedule for the assessment of Insight Scale Expanded version- SAI-E [Mean (Inter-Quartile Range); unit: units on a scale] — The Schedule for the assessment of Insight Scale Expanded version- SAI-E is a scale that measures insight as a multidimensional concept; including awareness of having a mental illness, ability to relabel psychotic phenomena as abnormal and compliance with treatment. The score is between 1 and 35. The higher score represents a better insight.
  units on a scale | 12.4 [7.0 to 18.3] | 15.0 [8.9 to 21.0] | 14.0 [7.8 to 19.8]
First domain (physical health) of The World Health Organization Quality of Life WHOQOL-BREF [Mean (Standard Deviation); unit: units on a scale] — First domain (physical health) of The World Health Organization Quality of Life WHOQOL- BREF which is a short form of the World Health Organization Quality of Life scale. The minimum score is 0 and the highest is 100. The higher the score the better quality of life.
  units on a scale | 62.4 (16.1) | 63.5 (15.9) | 62.9 (15.9)
Second domain (psychological) of The World Health Organization Quality of Life WHOQOL-BREF [Mean (Standard Deviation); unit: units on a scale] — Second domain (psychological) of The World Health Organization Quality of Life WHOQOL-BREF which is a short form of the World Health Organization Quality of Life scale. The minimum score is 0 and the highest is 100. The higher the score the better quality of life.
  units on a scale | 61.5 (16.6) | 61.4 (17.8) | 61.5 (17.2)
Third domain (social relationships) of The World Health Organization Quality of Life WHOQOL-BREF [Mean (Standard Deviation); unit: units on a scale] — Third domain (social relationships) of The World Health Organization Quality of Life WHOQOL-BREF which is a short form of the World Health Organization Quality of Life scale. The minimum score is 0 and the highest is 100. The higher the score the better quality of life.
  units on a scale | 52.1 (21.2) | 53.2 (24.3) | 52.7 (22.7)
Fourth domain (environment) of The World Health Organization Quality of Life WHOQOL-BREF [Mean (Standard Deviation); unit: units on a scale] — Fourth domain (environment) of The World Health Organization Quality of Life WHOQOL-BREF which is a short form of the World Health Organization Quality of Life scale. The minimum score is 0 and the highest is 100. The higher the score the better quality of life.
  units on a scale | 61.7 (15.3) | 66.9 (13.7) | 64.3 (14.7)
Family Emotional Involvement and criticism Scale (FEICS) [Mean (Standard Deviation); unit: units on a scale] — Family Emotional Involvement and criticism Scale (FEICS) is a self-report scale to measure expressed emotion. The minimum value is 14 and the maximum value is 70. The higher the score the better expressed emotions.
  units on a scale | 29.6 (8.9) | 29.3 (8.6) | 29.5 (8.8)
Objective domain of the Family burden self-administered scale [Mean (Standard Deviation); unit: units on a scale] — Objective domain of the family burden self-administered scale is a scale for assessing caregiver burden. The minimum score is 0 and the maximum score is 2. The higher the score the more family burden.
  units on a scale | 0.44 (0.47) | 0.46 (0.44) | 0.45 (0.46)
Subjective domain of the family burden self-administered scale [Mean (Standard Deviation); unit: units on a scale] — Subjective domain of the family burden self-administered scale is a scale for assessing caregiver burden. The minimum score is 0 and the maximum score is 2. The higher the score the more burden.
  units on a scale | 0.92 (0.42) | 0.91 (0.45) | 0.92 (0.44)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Relapse
Description: Defined as the reappearance of criteria for an episode of psychosis in a patient who did not or only had residual symptoms. It can be set in two ways: hospitalization or a score on the CGI-S greater than or equal to 3 in the evaluation and an increase greater than 20% in the Scale for the Assessment of Positive Symptoms (SAPS)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Group Psychoeducation | Treatment as Usual Only
Number analyzed (Participants) | 90 | 86
Participants | 22 | 23
Statistical Analysis 1: Comparison: Brief Group Psychoeducation vs Treatment as Usual Only; Test type: Superiority; p = 0.59, Mixed Models Analysis; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.77 to 1.16] — This is intention-to-treat analysis. The Brief Group Psychoeducation is the numerator and the group of Treatment as Usual Only is the denominator for relative risk

2. Secondary Outcome: Number of Patients With Hospitalization
Description: Need confinement in a hospital or clinic.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Group Psychoeducation | Treatment as Usual Only
Number analyzed (Participants) | 90 | 86
Participants | 10 | 9
Statistical Analysis 1: Comparison: Brief Group Psychoeducation vs Treatment as Usual Only; Test type: Superiority; p = 0.73, Mixed Models Analysis; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.87 to 1.10] — The Brief Group Psychoeducation is the numerator and the group of Treatment as Usual Only is the denominator for relative risk. This is intention-to-treat analysis

3. Secondary Outcome: Symptoms of Schizophrenia
Description: Will be measured with rating Scales for the Assessment of Positive Symptoms (SAPS) and negative symptoms (SANS). The Scale for the Assessment of Positive Symptoms (SAPS) is a rating scale to measure positive symptoms in schizophrenia. SAPS is split into 4 domains, and within each domain separate symptoms are rated from 0 (absent) to 5 (severe). The score is between 0 and 155, a higher score on the scale represents a worse clinical status.The Scale for the Assessment of Negative Symptoms (SANS) is a rating scale to measure negative symptoms in schizophrenia. The scale is between 0 and 95. The higher score represents worse clinical status
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Group Psychoeducation | Treatment as Usual Only
Number analyzed (Participants) | 90 | 86
score on a scale
  SANS scale | 34.7 (18.4) | 35.6 (16.5)
  SAPS scale | 13.3 (17.6) | 10.9 (12.4)
Statistical Analysis 1: Comparison: Brief Group Psychoeducation vs Treatment as Usual Only; Test type: Superiority; p = 0.94, Mixed Models Analysis; Slope = 0.01, 95% CI 2-sided [-0.36 to 0.39] — This is intention-to-treat analysis
Statistical Analysis 2: Comparison: Brief Group Psychoeducation vs Treatment as Usual Only; Test type: Superiority; p = 0.30, Mixed Models Analysis; Slope = -0.19, 95% CI 2-sided [-0.57 to 0.18] — This is intention-to-treat analysis

4. Secondary Outcome: Adherence to Treatment
Description: Was defined in three categories: 1=Take regularly medication 100% of the time, 2 =Partial adherence 3= Does not take medication.
Time Frame: 12 months
Population: Data was not gathered for all the participants in this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Group Psychoeducation | Treatment as Usual Only
Number analyzed (Participants) | 63 | 52
Participants
  Takes regularly medication | 41 | 36
  Partial adherence | 21 | 16
  Does not take medication | 1 | 0

5. Secondary Outcome: Insight
Description: The Schedule for the assessment of Insight Scale Expanded version- SAI-E is a scale that measures insight as a multidimensional concept; including awareness of having a mental illness, ability to relabel psychotic phenomena as abnormal and compliance with treatment. The score is between 1 and 35. The higher score represents a better insight.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Group Psychoeducation | Treatment as Usual Only
Number analyzed (Participants) | 90 | 86
score on a scale | 14.9 (6.9) | 16.4 (5.5)
Statistical Analysis 1: Comparison: Brief Group Psychoeducation vs Treatment as Usual Only; Test type: Superiority; p = 0.61, Mixed Models Analysis; Slope = 0.03, 95% CI 2-sided [-0.10 to 0.17] — This is an intention to treat analysis

6. Secondary Outcome: Quality of Life Measure by WHOQOL-BREF
Description: First domain (physical health) of The World Health Organization Quality of Life WHOQOL- BREF which is a short form of the World Health Organization Quality of Life scale. The minimum score is 0 and the highest is 100. The higher the score the better quality of life. Second domain (psychological) the minimum score is 0 and the highest is 100. The higher the score the better quality of life.Third domain (social relationships) the minimum score is 0 and the highest is 100. The higher the score the better quality of life. Fourth domain (environment) the minimum score is 0 and the highest is 100. The higher the score the better quality of life.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Group Psychoeducation | Treatment as Usual Only
Number analyzed (Participants) | 90 | 86
score on a scale
  WHOQOL-BREF 1ST DOMAIN | 61.8 (14.0) | 63.6 (15.2)
  WHOQOL-BREF 2ND DOMAIN | 61.9 (16.4) | 62.6 (16.4)
  WHOQOL-BREF 3RD DOMAIN | 58.1 (17.7) | 57.8 (23.0)
  WHOQOL-BREF 4TH DOMAIN | 62.5 (13.9) | 65.8 (14.5)
Statistical Analysis 1: Comparison: Brief Group Psychoeducation vs Treatment as Usual Only; Test type: Superiority — This statistical Analysis applies to WHOQOL-BREF 1ST DOMAIN (physical health) in the first row; p = 0.81, Mixed Models Analysis; Slope = 0.04, 95% CI 2-sided [-0.38 to 0.30] — This is an intention to treat analysis. This statistical Analysis applies to WHOQOL-BREF 1ST DOMAIN (physical health) in the first row
Statistical Analysis 2: Comparison: Brief Group Psychoeducation vs Treatment as Usual Only; Test type: Superiority — This is an intention to treat analysis. This statistical Analysis applies to WHOQOL-BREF 2ND DOMAIN (psychological) in the second row; p = 0.81, Mixed Models Analysis; Slope = -0.04, 95% CI 2-sided [-0.38 to 0.29] — This is an intention to treat analysis.This statistical Analysis applies to WHOQOL-BREF 2ND DOMAIN (psychological) in the second row
Statistical Analysis 3: Comparison: Brief Group Psychoeducation vs Treatment as Usual Only; Test type: Superiority — This statistical Analysis applies to WHOQOL-BREF 3RD DOMAIN (social relationships) in the third row; p = 0.52, Mixed Models Analysis; Slope = 0.16, 95% CI 2-sided [-0.33 to 0.65] — This is an intention to treat analysis. This statistical Analysis applies to WHOQOL-BREF 3RD DOMAIN (social relationships) in the third row
Statistical Analysis 4: Comparison: Brief Group Psychoeducation vs Treatment as Usual Only; Test type: Superiority — This statistical Analysis applies to WHOQOL-BREF 4TH DOMAIN (environment) in the fourth row; p = 0.27, Mixed Models Analysis; Slope = 0.19, 95% CI 2-sided [-0.15 to 0.53] — This is an intention to treat analysis. This statistical Analysis applies to WHOQOL-BREF 4TH DOMAIN (environment) in the fourth row

7. Secondary Outcome: Family Burden
Description: Is defined as the impact it may have on the caregiver who lives with a psychiatric patient. It is evaluated with the Self-Administered Scale of Family Burden (SSFB) which has 2 domains: Objective domain measures the alterations of daily behavior of the patients family. The minimum score is 0 and the maximum score is 2. The higher the score the more family burden. Subjective domain is the stress produced by the patients behavior to the family. The minimum score is 0 and the maximum score is 2. The higher the score the more burden.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Group Psychoeducation | Treatment as Usual Only
Number analyzed (Participants) | 90 | 86
score on a scale
  SSFB objective domain | 0.66 (0.40) | 0.68 (0.37)
  SSFB subjective domain | 0.69 (0.37) | 0.76 (0.34)
Statistical Analysis 1: Comparison: Brief Group Psychoeducation vs Treatment as Usual Only; Test type: Superiority — This analysis applies to SSFB objective domain in the first row; p = 0.33, Mixed Models Analysis; Slope = -0.01, 95% CI 2-sided [-0.01 to 0.01] — This is an intention to treat analysis. This analysis applies to SSFB objective domain in the first row
Statistical Analysis 2: Comparison: Brief Group Psychoeducation vs Treatment as Usual Only; Test type: Superiority — This is an intention to treat analysis. This analysis applies to SSFB subjective domain in the second row; p = 0.19, Mixed Models Analysis; Slope = -0.01, 95% CI 2-sided [-0.02 to 0.01] — This is an intention to treat analysis. This analysis applies to SSFB subjective domain in the second row

8. Secondary Outcome: Expressed Emotions
Description: Are the attitudes of family members that interfere in interpersonal relations and it has shown to influence the course of psychiatric disorders, increasing the risk of relapse. The most studied are criticism and emotional over involvement. The first one is a negative filter that distorts the perceptions of a person over others. Over involvement is a lack of appropriate emotional limits among members of a family. They will be evaluated with the Family Emotional Involvement and Criticism Scale (FEICS). The minimum value is 14 and the maximum value is 70. The higher the score the better expressed emotions.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brief Group Psychoeducation | Treatment as Usual Only
Number analyzed (Participants) | 90 | 86
score on a scale | 31.1 (5.4) | 30.8 (6.6)
Statistical Analysis 1: Comparison: Brief Group Psychoeducation vs Treatment as Usual Only; Test type: Superiority; p = 0.97, Mixed Models Analysis; Slope = 0.01, 95% CI 2-sided [-0.19 to 0.19] — This is an intention to treat analysis

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Brief Group Psychoeducation | Treatment as Usual Only
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/86
Other Adverse Events (participants affected / at risk) | 0/90 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No